CLINICAL TRIAL: NCT06766110
Title: Evaluation of Upper Extremity Functions in Patients with Obesity Hypoventilation Syndrome
Brief Title: Evaluation of Upper Extremity Functions in Obesity Hypoventilation Syndrome Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Nilgün Yıldız, Physiotherapist, Istanbul University - Cerrahpasa
Other Study IDs: IUC-FTR-NYildiz-01
Record Dates: First submitted 2025-01-03; First posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Obesity Hypoventilation Syndrome (OHS)
Keywords: Obesity Hypoventilation Syndrome (OHS); upper extremity function; hand grip strength; activities of daily living
MeSH Terms: conditions — Obesity Hypoventilation Syndrome | interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Subjects with Obesity Hypoventilation Syndrome
  Interventions: Other: Assessment

INTERVENTIONS:
Other: Assessment — 31 volunteer participants who were followed up at the Department of Chest Diseases, Istanbul University, Istanbul Faculty of Medicine and met the inclusion criteria were included in the study. Participants' body composition, upper extremity functional exercise capacity, grip strength, and activities of daily living were evaluated.

SUMMARY:
Obesity Hypoventilation Syndrome (OHS) is a disease characterized by daytime hypercapnia and sleep-related respiratory disturbances in individuals with a body mass index (BMI) greater than 30 kg/m², without any other condition that could lead to hypoventilation. Although various mechanisms play a role in the pathogenesis of OHS, the most significant one is the altered respiratory system mechanics due to obesity. Obesity also leads to a decrease in peripheral muscle strength and exercise capacity. It has been reported that in obese individuals, not only general body movements and lower extremities but also upper extremity movements are negatively affected. Specifically, it has been observed that during activities against gravity, movement speed is low while the duration of movement is high. In OHS patients, daily living activities, physical activity, and exercise capacity are also negatively impacted. Supported or unsupported arm movements are of great importance in performing daily living activities. The muscles activated during both simple arm lifting and combined movements also function as accessory respiratory muscles. In individuals with cardiopulmonary diseases, an increase in the respiratory workload, especially during unsupported arm movements, has been observed. It is thought that in OHS patients, both the effects of obesity and the respiratory system may limit upper extremity functions. However, no studies have evaluated upper extremity functions in these individuals. Therefore, the aim of investigators study is to evaluate upper extremity functions in OHS patients.

DETAILED DESCRIPTION:
The study will include patients diagnosed with Obesity Hypoventilation Syndrome, who are followed at the Department of Chest Diseases, Istanbul University Faculty of Medicine. The study will be conducted in accordance with the Helsinki Declaration, and an informed consent form will be obtained from the participants who are willing to take part in the study. Before the study begins, the participants will be informed about the purpose of the study and provided with all relevant details. Participants who agree to participate will be invited to the Chest Diseases Department of Istanbul University Faculty of Medicine. Demographic information of the participants will be recorded, followed by the evaluation of body composition, upper extremity functional exercise capacity, grip strength, and activities of daily living. The main aim of the study is to comprehensively investigate the upper extremity functions in patients with OHS.

ELIGIBILITY:
Inclusion Criteria:

* Individuals between the ages of 18-65
* Individuals diagnosed with OHS by a Chest Disease Specialist

Exclusion Criteria:

* Individuals with neurological or orthopedic problems that prevent them from performing the tests or understanding the scales applied within the scope of the study
* Additional pulmonary disease
* Uncontrolled cardiovascular disease
* Presence of uncontrolled diabetes

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with Obesity Hypoventilation Syndrome who are followed up at the Department of Chest Diseases of Istanbul University Istanbul Faculty of Medicine will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
6-Minute Pegboard and Ring Test - Upper Extremity Functional Exercise Capacity | 1 day
  For the test, a perforated wooden board and bars, adjustable according to shoulder levels, are used. The participant sits in front of the board, which has a total of four sticks: two placed at shoulder level and shoulder width, and two placed 20 cm above this level. Ten rings are placed on the lower sticks. The participant is instructed to use both hands simultaneously to move the rings from the lower stick to the upper one and return them to the lower stick once completed. They are asked to perform this task as quickly as possible for 6 minutes. The number of rings is recorded and heart rate, blood pressure, oxygen saturation, fatigue, and dyspnea are measured before and after the test.
Milliken Activities of Daily Living Scale | 1 day
  This scale is a self-reported assessment that evaluates upper extremity dysfunctions and shows limitations in ADL. It consists of 6 sections: meal preparation and eating (8 items), personal hygiene (9 items), dressing (8 items), object manipulation (9 items), house cleaning (7 items), and other activities (6 items), totaling 47 items. For each item, both ability and requirement levels are scored; the ability level uses a 1-5 scale, and the requirement level uses a 1-3 scale.
Grip Strength | 1 day
  Grip strength is measured with a Jamar hand dynamometer recommended by the American Hand Therapists Association. Measurements are made with the participant in shoulder adduction, elbow 90° flexion, forearm neutral, and wrist 0-30° extension. The participant is asked to squeeze the dynamometer with maximum force and hold for 3 seconds. Measurements are repeated 3 times on the dominant and non-dominant hands, and the results are recorded in kg.
The Glittre Activities of Daily Living Test | 1 day
  The test starts from a seated position on a 10-meter surface. After walking 5 meters, the participant climbs a two-step ladder, walks to the shelves, and moves three 1 kg objects from the top shelf to the middle and bottom shelves, then returns them to the middle and top shelves. The participant then turns around, climbs the stairs, and sits back down. This completes one full round, and a total of 5 rounds are performed. The participant is asked to complete the rounds as quickly as possible. Women carry a 2.5 kg backpack, and men carry a 5 kg backpack. The completion time is recorded, and heart rate, blood pressure, oxygen saturation, fatigue, and dyspnea are measured before and after the test.

SECONDARY OUTCOMES:
Body Mass Index | 1 day
  Body mass index (BMI) is calculated by dividing body weight in kilograms (kg) by the square of height in meters (m). BMI is calculated from the formula body weight/height² (kg/m²).
Anthropometric Measurements - Waist Circumference | 1 day
  Waist circumference is measured in cm using a standard non-elastic tape measure from the midpoint between the subcostal region and the iliac crest after full expiration.
Anthropometric Measurements - Hip Circumference | 1 day
  Hip circumference is measured from the widest part of the hip, with the tape measure parallel to the floor.
Anthropometric Measurements - Neck Circumference | 1 day
  Neck circumference is measured horizontally from the lower border of the laryngeal prominence with the head in an upright position.
Anthropometric Measurements - Arm Circumference | 1 day
  Arm circumference is measured from the midpoint of the distance between the acromion and the olecranon, which is the most swollen part of the muscle.
The Waist-Hip Ratio | 1 day
  Waist and hip circumference will be measured in cm with the help of a tape measure. It is calculated by dividing the waist circumference by the hip circumference.
Body Fluid Percentage | 1 day
  Participants body fluid percentage will be measured using the 'Tanita BC-545N Body Analysis Scale' with the bioelectrical impedance analysis method.
Body Fat Percentage | 1 day
  Participants body fat percentages will be evaluated using the "Tanita BC-545N Body Analysis Scale" with the bioelectrical impedance analysis technique.
Muscle Mass | 1 day
  Participants' muscle mass will be assessed using the "Tanita BC-545N Body Analysis Scale" with the bioelectrical impedance analysis technique. The results will be recorded in kg.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided